CLINICAL TRIAL: NCT02524184
Title: Sildenafil Activates Browning of White Adipose and Improves Insulin Sensitivity in Human Adults
Brief Title: Sildenafil Activates Browning of White Adipose and Improves Insulin Sensitivity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wze20150088
Record Dates: First submitted 2015-08-02; First posted 2015-08-14 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Eleven patients receive sildenafil 100mg/day (25 mg at 8 AM plus 25 mg at 4 PM plus 50 mg at 10 PM)for 7 days.
  Interventions: Drug: sildenafil
- Placebo group (Placebo Comparator): An identical placebo for 7 days in placebo group.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sildenafil — sildenafil 100 mg per day for 7 days.
  Arms: Sildenafil
Drug: placebo — an identical placebo per day for 7 days
  Arms: Placebo group

SUMMARY:
Obesity and metabolic disease result when energy intake consistently exceeds energy expenditure. One appealing new target for treatment is the activation of brown adipose tissue (BAT), an organ recently found to be functional in adult humans. Brown adipocytes selectively express uncoupling protein 1 (UCP1), which renders the inner membrane of mitochondria leaky, thereby diverting chemical energy from ATP generation to heat production. Interest in BAT has been spurred by the recognition that in addition to classical BAT depots, other brown-fat-like cells are present in the subcutaneous white adipose tissue (WAT) in animals and also in humans.These cells have structural and functional properties that resemble brown adipocytes, and they are referred to as beige or 'brite' (brown-in-white) adipocytes. Interestingly, browning of WAT can be induced in animals and humans by physiological stimuli such as cold exposure, which increases adrenergic tone, and by exercise, which selectively drives WAT browning through irisin, an exercise-induced myokine. In addition b-adrenergic drugs and other pharmacological agents,such as prostaglandins, can induce browning of white adipose tissue. More recently, one study showed that treatment of C57BL/6 mice with phosphodiesterase inhibitor sildenafil (12 mg/kg/d) for 7 d caused 4.6-fold increase in uncoupling protein-1 expression and promoted establishment of a brown fat cell-like phenotype ("browning") of WAT in vivo. Therefore, the investigators hypothesized that sildenafil can promote browning of white adipose tissue and improves insulin sensitivity in human adults.

DETAILED DESCRIPTION:
The study subjects will be taken placebo (first stage) and sildenafil (second stage) intervention for 7 days, respectively afterward.Subcutaneous fat tissue and muscle samples will be obtained by biopsy from some individuals and measure the browning of white adipose tissue and insulin signaling.The insulin sensitivity will be tested by insulin clamp assay before and after each intervention, respectively. In addition,blood samples for biochemical analysis will be obtained before and after each intervention, respectively.

The browning of white adipose tissue will be measured by the expressions of peroxisome proliferator-activated receptor-γ (PPARγ), PPARγcoactivator 1α (PGC-1α), uncoupling protein 1 (UCP-1), the second messenger cyclic guanosine-3', 5'-monophosphate (cGMP),PR domain containing 16 zinc finger transcription factor (Prdm16) and deiodinase, iodothyronine, type II (DIO2).The metabolic makers will be measured by blood pressure, heart rate, thyroid functions, resting metabolic rate, respiratory quotient, blood cGMP, blood insulin and blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* overweight volunteers
* 20-30 years old
* body mass index >=25 kg/m2
* normal glucose tolerance

Exclusion Criteria:

* normal body mass index
* abnormal cardiovascular status
* women
* history of any local or systemic infectious disease with fever or requiring antibiotic within four weeks of drug administration
* current addiction to alcohol or substances of abuse
* children
* current addiction to alcohol or substances of abuse
* mental incapacity
* the use of any medication within four weeks
* subjects with hyperthyroidism or hypothyroidism, hypertension (even if controlled with medications)

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Browning of white adipose tissue | 7 days
  The browning of white adipose tissue was measured by Western blot (including the expressions of peroxisome proliferator-activated receptor-γ (PPARγ), PPARγcoactivator 1α (PGC-1α), uncoupling protein 1 (UCP-1), the second messenger cyclic guanosine-3', 5'-monophosphate (cGMP),PR domain containing 16 zinc finger transcription factor (Prdm16) and deiodinase, iodothyronine, type II (DIO2)).

SECONDARY OUTCOMES:
Improvement of insulin sensitivity | 7days
  The insulin sensitivity will be tested by insulin clamp before and after each intervention,respectively.

OTHER OUTCOMES:
Change of metabolic status | 3 months
  The metabolic status including blood pressure, heart rate, thyroid functions, resting metabolic rate, respiratory quotient, blood cGMP, blood insulin and blood glucose will be measured before and after intervention in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan General Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Li S, Li Y, Xiang L, Dong J, Liu M, Xiang G. Sildenafil induces browning of subcutaneous white adipose tissue in overweight adults. Metabolism. 2018 Jan;78:106-117. doi: 10.1016/j.metabol.2017.09.008. Epub 2017 Oct 3. PMID 28986166